CLINICAL TRIAL: NCT06661499
Title: An Observational Clinical Study on the Construction of an Artificial Neural Network Model for Rapid Intelligent Diagnosis of Microorganisms in ICU Pneumonia Based on Species-specific Rapid Detection of Pathogenic Bacteria
Brief Title: An Observational Clinical Study on the Construction of an Artificial Neural Network Model for ICU Pneumonia
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: 2024-607-01
Record Dates: First submitted 2024-09-05; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-08

CONDITIONS: Pneumonia
Keywords: pneumonia; colonization; infection; artificial neural network model; intensive care unit
MeSH Terms: conditions — Pneumonia; Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: establish an artificial neural network model — to establish an artificial neural network model for pathogen diagnosis in ICU pneumonia

SUMMARY:
To achieve rapid, intelligent and accurate microbiological diagnosis and treatment for ICU pneumonia, an artificial neural network model for microbiological diagnosis is established, which depends on many clinical cases and machine deep learning from clinical experts' judgements according to species-specific rapid detection of pathogenic bacteria and other clinical parameter variables of patients.

DETAILED DESCRIPTION:
This study is a prospective single-centre observational study, 600 ICU pneumonia patients are expected to be selected as the observation object, and the lower respiratory secretions of patients on d1, d3 and d7 after enrollment are collected for species-specific rapid detection and microbial culture, while the general information of the patients and the clinical information of the corresponding time points on d1, d3 and d7 are collected. Two experienced senior physicians were organized to determine whether the microbial results were colonized or infected, and an artificial neural network model for rapid and intelligent diagnosis of pathogenic microorganisms in ICU pneumonia will be established and validated through multi-dimensional machine learning.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥18 years;
2. agreed to obtain lower respiratory specimens for rapid testing of pathogenic bacteria;
3. all were enrolled by an experienced physician who dynamically determined that the microorganisms were in a colonised or infected state;
4. signed an informed consent form.

Exclusion Criteria:

1. pregnant women;
2. lactating women;
3. patients who could not obtain lower respiratory specimens;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pneumonia patients who admitted to Nanjing Drum Tower Hospital from Jan 1,2025 to Dec 31,2027 and meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
clinical evaluation of each microbial detected whether in colonization or infection | day1,day3 and day7 after enrollment
  Two experienced senior physicians are organized to determine whether the microbial are colonized or infected according to clinical values.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Master, Principal Investigator — Nanjing Drum Tower Hosptial
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No